CLINICAL TRIAL: NCT02364908
Title: Prospective Evaluation of Adherence to Antimalarials in Patients With Systemic Lupus and Role of Therapeutic Education
Brief Title: Prospective Evaluation of Decision and Compliance With Antimalarials in Patients With Systemic Lupus
Acronym: ESSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Région Nord-Pas de Calais, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013_65; 2014-A00735-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: systemic lupus erythematosus; antimalarials; therapeutic education; Coping questionnaire; MASRI questionnaire; morisky medication adherence scale; lupus Quality Of Life; internal medicine
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Systemic Lupus (Other)
  Interventions: Other: therapeutic education

INTERVENTIONS:
Other: therapeutic education — This is the group sessions aimed to convey additional information to patients about their disease. The main objective is to learn how to better anticipate any medical problems and better manage daily life with the disease.

SUMMARY:
This study is a biomedical, open label, therapeutic strategy, interventional, non-randomized, multicenter study to evaluate the non compliance to antimalarials in patients with systemic lupus in the Nord Pas-de-Calais region (FRANCE). It is conducted in two visits. These visits consist in obtaining blood sample, performing a clinical examination and filling in a questionnaire (Quality Of Life, Coping...).

The goal for the noncompliants patients is to guide them towards the therapeutic education with professionals (nurses and physicians).

ELIGIBILITY:
Inclusion Criteria:

* patients with a systemic lupus with ACR criteria (at least 4 criterias)
* patients with antimalarials for at least 3 months with a minimum dose of 200 mg/day.

Exclusion Criteria:

* patients who refuse to sign the informed consent
* patients who are under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
measure of the frequency of patients with systemic lupus noncompliants to their antimalarials treatment. | baseline, at 12 months

SECONDARY OUTCOMES:
hydroxychloroquinémie | between 6 months at 12 months
  Monitoring of blood levels of hydroxychloroquinémie
number of non- adherent patients | at 12 months
  Identification of the number of non- adherent patients are being enrolled in Education Protocol Patient and number of sessions followed ;
quality of life scale Coping | baseline, at 12 months
  scale Coping ( WCC-R Par COUSSON et al. (1996) ) scale MASRI, scale MMAS-8-item

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hachulla, MD, PhD, Study Chair — University Hospital, Lille
Locations (7):
- France (7):
  - CH Hôpital Duchenne, Boulogne-sur-Mer
  - CH Douai, Douai
  - CH Dunkerque, Dunkirk
  - CH du Dr Schaffner, Lens
  - CHRU, Hôpital Huriez, Lille
  - Victor Provo Hospital, Roubaix
  - Valenciennes hospital, Valenciennes

IPD SHARING:
Plan to Share IPD: No